CLINICAL TRIAL: NCT06150430
Title: An Active Pelvis Orthosis (APO) for Post-stroke Gait Rehabilitation: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IUVO S.r.l. (Industry)
Collaborators: Össur Iceland ehf (Industry); Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ortesi_Pelvica_Attiva_02
Record Dates: First submitted 2023-11-13; First posted 2023-11-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: Hip exoskeleton; Cerebrovascular Disorders; Nervous System Diseases
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Training with APO (Experimental): All participants are assigned to the training group with the APO
  Interventions: Device: APO

INTERVENTIONS:
Device: APO — Subjects will take part in 14 experimental sessions: two baseline sessions (T1-T2), three familiarization sessions (F1-F3), six training sessions (E1-E6), two assessment sessions (one pre-training T3 and one post training T4) and one 2-month follow-up session (T5). Depending on the session, the subject will walk with and/or without the APO. During the assessment sessions (T3-T4), the subject will be evaluated through different standard tests (such as 10MWTs and 2mWTs) and instrumented gait analysis, with and without the APO.
  The goal of each training session (E1-E6) will be to achieve a minimum of 30 minutes of overground walking assisted by the APO, leaving up to 15 minutes to rest if needed. Training sessions will occur 2-3 times a week for 2-3 weeks to complete the training protocol.

SUMMARY:
The primary objective of this study is to evaluate the safety, reliability and short-term effectiveness of APO-based training to increase the self-selected walking velocity (SSV) of stroke patients. The robotic device is the Active Pelvic Orthosis RT v3.1 (IUVO APO) developed bu IUVO S.r.l.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety, reliability and short-term effectiveness of APO-based training to increase the self-selected walking velocity (SSV) of stroke patients. The endpoint to evaluate the APO-based training effectiveness will be the difference in self-selected walking velocity (m/s) comparing post-training session (T4) to baseline sessions (T1&T2).

Other objective of the study, both secondary and exploratory, have been defined to further investigate the effects of the IUVO APO on post-stroke subjects.

The Investigational Device, Active Pelvis Orthosis RT v3.1 (APO), is a bilateral powered robotic hip orthosis (or exoskeleton) designed to gently assist hip flexion-extension movements by providing smooth assistive torque at the hip level, automatically adapting to natural gait variations.

The study will be an interventional single-arm clinical trial with no control group and will involve up to 20 subjects, that fulfil the inclusion/exclusion criteria. This should be sufficient to provide the input needed to reach the primary and secondary objectives of the trial.

In the protocol, after the screening visit, subjects will take part in 14 experimental sessions: two baseline sessions (T1-T2), three familiarization sessions (F1-F3), six training sessions (E1-E6), two assessment sessions (one pre-training T3 and one post training T4) and one 2-month follow-up session (T5). Depending on the session, the subject will be asked to walk with or without the APO, or both. During the assessment sessions, the subject will be evaluated through different standard tests (such as 10MWTs and 2mWTs) and instrumented gait analysis, with and without APO. In the training sessions, the subject will perform some overground walking practice with APO.

ELIGIBILITY:
Inclusion Criteria:

* cerebral stroke;
* at least 3 months from cerebral event;
* hemiparesis;
* age > 18 years;
* SSV greater than 0.3 (m/s);
* SSV less than 0.8 (m/s);
* ability to ambulate with no more than minimal contact assistance;
* maximum hip width range, i.e., distance between Great Trochanters = 430 mm.

Exclusion Criteria:

* Modified Ashworth Scale >3 at the hip and/or ankle joints;
* inability to follow verbal 3 step commands;
* severe aphasia causing inability to communicate with the investigators;
* serious medical conditions (recent myocardial infarction in less than 3 months, uncontrolled congestive heart failure (CHF), uncontrolled hypertension, uncontrolled seizures);
* leg deep vein thrombosis less than 6 weeks ago;
* other pre-existing neurological disorders (Parkinson's disease, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Dementia);
* Severe osteoporosis;
* severe hip / knee osteoarthritis with limitation of movement or significant pain;
* use of a colostomy bag;
* skin wounds, infection or problems at device contact locations;
* major orthopedic surgery or fractures within the last 90 days (hip, knee, ankle, foot, spine);
* cardiac surgery within the last 3 months;
* patient has recently or is currently participating in research that may influence, in PI's opinion, responses to study intervention;
* pregnancy;
* breastfeeding woman;
* implanted cardiac devices (pacemakers, ICDs);
* use of assistive device that, in the PI's opinion, could interfere with APO;
* it is recommended that participants treated with anti-spasticity agents (oral, injectable or intrathecal) keep the dosage for these medications constant throughout the study;
* where medically appropriate, all other concomitant medications being taken by a participant at entry into the study should continue at the same dose until end of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Device Events (ADEs) and Serious Adverse Device Events (SADEs) | Duration of the study participation (estimated 4 weeks, excluding follow-up)
  Safety of the device will be assessed by the number of ADEs and SADEs throughout the duration of the study
Incidence of Adverse Device Events (ADEs), Serious Adverse Device Events (SADEs) and Device Deficiencies (DDs) | Duration of the study participation (estimated 4 weeks, excluding follow-up)
  Reliability of the device will be assessed by the number of ADEs, SADEs and DDs throughout the duration of the study
10-Meter Walk Test (10MWT) at Self-Selected walking Velocity (SSV) | Baseline, Post-Training (estimated 3-4 weeks)
  Change in SSV measured without the device

SECONDARY OUTCOMES:
10-Meter Walk Test (10MWT) at Fast walking Velocity (FV) | Baseline, Post-Training (estimated 3-4 weeks)
  Change in FV measured without the device
10-Meter Walk Test (10MWT) at Self-Selected walking Velocity (SSV) | Post-Training (estimated 3-4 weeks), Follow-up (2 months follow up)
  Change in SSV measured without the device
10-Meter Walk Test (10MWT) at Fast walking Velocity (FV) | Post-Training (estimated 3-4 weeks), Follow-up (2 months follow up)
  Change in FV measured without the device
2-minute Walk Test (2mWT) | Baseline, Post-Training (estimated 3-4 weeks)
  Change in walking endurance measured without the device
2-minute Walk Test (2mWT) | Post-Training (estimated 3-4 weeks), Follow-up (2 months follow up)
  Change in walking endurance measured without the device

CONTACTS AND LOCATIONS:
Overall Officials: Franco Molteni, MD, Principal Investigator — Ente Ospedaliero Valduce - UOC di Medicina Riabilitativa Villa Beretta
Locations (1):
- Ente Ospedaliero Valduce - UOC di Medicina Riabilitativa Villa Beretta, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No